CLINICAL TRIAL: NCT05759806
Title: Safety and Performance Evaluation of the Nephronyx System for the Treatment of Patients With ADHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nephronyx LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-NPX-085
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Acute Decompensated Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADHF patients (Experimental): ADHF patients with compromised response to diuretics treated with Nephronyx system
  Interventions: Device: Nephronyx system (Perfuser)

INTERVENTIONS:
Device: Nephronyx system (Perfuser) — Temporary deployment of the Nephronyx system (Perfuser)
  Other Names: The Nephronyx system (Perfuser)

SUMMARY:
The objective of this interventional study is to evaluate the safety and functional performance of the Nephronyx System in patients with ADHF, presenting clinical signs of volume overload and compromised response to diuretics.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the hospital with a primary diagnosis of ADHF
* Patient has signs of volume overload as evidence by a score of ≥ 4 on the EVEREST score
* Patient with Left Ventricular Ejection Fraction LVEF >15%
* Patient has compromised response to diuretics
* NT-proBNP >450 pg/mL if aged <55 years, >900 pg/mL if aged between 55 and 75 years and >1800 pg/mL if aged >75 years

Exclusion Criteria:

* Patient with active DVT or history of DVT
* Patient has documented or evidence of Renal artery stenosis
* BMI>35 Kg/m^2
* Patient has documented, untreated symptomatic coronary artery disease (CAD) requiring revascularization
* Patient is in Cardiogenic shock
* Patient has blood dyscrasia, acute anemia, thrombocytopenia, bleeding diathesis, or coagulopathy
* Temperature > 38°C, or sepsis, or active systemic infection requiring IV anti-microbial treatment
* Patient has shown liver cirrhosis or has signs of liver damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 24 hours post device retrieval
  Device and/or investigational procedure related SAEs
Performance/ Procedural success | procedure day
  Device preforms as planned with no associated device malfunction

CONTACTS AND LOCATIONS:
Overall Officials: Doron Aronson, MD, Study Director — Rambam Health Care Campus
Locations (4):
- Israel (4):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - The Baruch Padeh Medical Center, Poriya, Poria Illit
  - Kaplan Medical Center, Rehovot

IPD SHARING:
Plan to Share IPD: No